CLINICAL TRIAL: NCT05015218
Title: Internal Jugular Vein Ultrasound for the Prediction of Spinal-induced Hypotension in Dehydrated Elderly Patients With Orthopaedic Trauma
Brief Title: Internal Jugular Vein and Spinal-induced Hypotension
Status: Completed | Type: Observational
Sponsor: Attikon Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, THEODOSIOS SARANTEAS, Professor, Attikon Hospital
Other Study IDs: ID: EBΔ 630 (23/11/2021)
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Haemodynamic Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vacular Ultrasound — To visualize the internal jugular veins ( IJVs) a linear transducer with a 5-10 MHz linear probe was placed over the neck, and the IJV was measured just below the bifurcation of the sternal and clavicular heads of the muscle. The IJV measurements were performed on the transverse axis over a single respiratory cycle. Patients with evidence of IJV thrombosis were excluded. IJV measurements included the antero-posterior maximum diameter at the end of expiration (IJVmax), the antero-posterior mimimum diameter/area at the end of inspiration (IJVmin), the IJV collapsibility index (IJV-CI) during spontaneous, quiet, breathing, [(IJVmax - IJVmin area)/IJVmax] and the ratio (R) of IJVmax-to-IJV-CI.
  Other Names: Blood pressure recordings

SUMMARY:
The study aims to assess internal jugular vein ultrasound derived measurements and indices prior to spinal anesthesia in elderly population who fulfills predetermined inclusion criteria and might greatly benefit from an appropriate hemodynamic control during orthopedic surgery. Therefore, it is evaluated the diagnostic performance of these indices in predicting spinal-induced hypotension in this subset of participants.

DETAILED DESCRIPTION:
Study design; Observational

1. Recruitment: Preoperative anesthetic and cardiovascular evaluation by the anesthesiology department as well as the cardiology department to define patients with predetermined criteria. Patients' medical history, blood tests (e.g. blood urea and cratinine) physical examination, electrocardiogram (ECG), and X-ray assessment are performed during the pre-operative assessment, supplemented by specific exams or tests (e.g. TTE, troponin or pro-BNP levels) as per the consultant cardiologists' recommendations.

   Consecutive sampling of aging patients (>70 years), who sustain trauma of the lower limb(hip fractures) undergoing an orthopedic surgical procedure (hip fracture repair) and planned spinal anesthesia. More specifically, patients included, are subjected to an orthopaedic surgical repair of a proximal femur fracture under spinal anaesthesia. All patients or their relatives provide a written consent to participate in the study.
2. Inclusion criteria/initial screening: Age>70 years. Nitrogen Urea/Creatinine>20.American College of Cardiology (ACC) stage I or II.

Exclusion criteria includes severe pulmonary hypertension/tricuspid regurgitation, tachycardia (heart rate > 100 beats/min), atrial fibrillation. Additionally, all patients who has spinal anaesthesia and the maximum cephalad dermatomal extension of the sensory block is below T12 are excluded from the study. Arterial hypotension related to overt intra-operative bleeding (>150 cc) or patients requiring blood transfusion, for any reason, is not considered in the statistical analysis.

2. Preoperative POCUS IJV ultrasonography To visualize both the right and left IJV a linear transducer with a 5-10 MHz linear probe is placed over the neck, and the IJV is measured just below the bifurcation of the sternal and clavicular heads of the muscle. The IJV measurements are performed on the transverse axis during spontaneous quiet, breathing. Patients with evidence of IJV thrombosis are excluded. IJV measurements included the maximum area at the end of expiration (IJVmax), the minimum area at the end of inspiration (IJVmin), the IJV collapsibility index (IJV-CI): [(IJVmax - IJVmin area)/IJVmax] and the ratio (R) of IJVmax-to-IJV-CI. Two examiners each performed all the measurements, generating two values; the mean of these values is used for analysis.

3. Anesthetic protocol and measurements. Spinal anesthesia is introduced with a single intrathecal injection of 0.75% (15 mg) plain ropivacaine using a 22 or 25-gauge needle with the patient in the lateral or sitting position. Intraoperative ECG, SPO2 and non-invasive blood pressure (measurements every two minutes) monitoring are routinely used. The non-invasive blood pressure is measured every 2 minutes and vital parameters are recorded continuously throughout surgery.

Patients experiencing a MAP (two consecutive measurements) less than or equal to 65 mmHg, or greater than or equal to 25% reduction of its baseline preoperative value is considered hypotensive Arterial hypotension related to bone cement application, intraoperative/postoperative bleeding with blood loss greater than 150cc or patients receiving blood transfusion for any reason are not considered in our statistical analysis.

The degree of sensory block (cold test) is assessed by an anesthesia staff not further involved in the study.

4. Follow up: Assessing hypotension due to spinal-anesthesia intraoperatively.

4. Statistical analysis Sample size: Previously, many echocardiographic indices have been used to predict spinal-induced hypotension. The collapsibility index of the inferior vena cava has showed an area under the curve in a receiver operating characteristic curve analysis between 0.77. We hypothesized, therefore, that the area under the curve of the IJV-CI would be at least 0.77 to predict spinal induced hypotension. We calculated the required sample size for the comparison of the area under a receiver operating characteristic curve with a null hypothesis value. Considering the α error of 0.05 with 90% power, 42 patients are needed. To allow for a possible 20% dropout rate, at least a sample size of 50 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Dehydrated elderly patients with orthopaedic trauma of the lower limb,
2. American Heart Association/American College of Cardiology (ACC) stage I or II.
3. Cardiac disease is in a compensated status.

Exclusion Criteria:

1. Atria fibrilation/Tachycardia (heart rate > 100 beats/min)
2. Sensory block less than T12
3. Overt intraoperative bleeding
4. Severe pulmonary hypertensopn/tricuspid regurgitation

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Consecutive sampling is used to recruit dehydrated aging patients (>70 years), who sustain trauma of the lower limb and underwent an orthopedic surgical procedure under spinal anesthesia.
  Patients' medical history, blood tests, physical examination, ECG, and X-ray assessment are standard practice, supplemented by specific exams or tests (e.g. TTE or pro-BNP levels), were performed per the consultant cardiologist's recommendations. All patients in our study were American Heart Association/American College of Cardiology (ACC) stage I, II and their cardiac disease is in a compensated status;
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Internal jugular vein aerea (cm2) prior to spinal anesthesia implementation | 10 minutes prior to spinal anesthesia
  Using GE-T8 Ultrasound System device, the right and leftinternal jugular vein is visualized on the short axis with a 5-10 MHz linear probe in B-mode.

CONTACTS AND LOCATIONS:
Overall Officials: HEODOSIOS SARANTEAS, PROFESSOR, Principal Investigator — MEDICAL SCHOOL UNIVERSITY OF ATHENS, NKUA, GREECE
Locations (2):
- Greece (2):
  - Department of anesthesia ,ATTIKON UNIVERSITY HOSPITAL OF ATHENS, Athens, Attica
  - Theodosios Saranteas, Athens, Gerakas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saranteas T, Spiliotaki H, Koliantzaki I, Koutsomanolis D, Kopanaki E, Papadimos T, Kostopanagiotou G. The Utility of Echocardiography for the Prediction of Spinal-Induced Hypotension in Elderly Patients: Inferior Vena Cava Assessment Is a Key Player. J Cardiothorac Vasc Anesth. 2019 Sep;33(9):2421-2427. doi: 10.1053/j.jvca.2019.02.032. Epub 2019 Feb 22. PMID 30904260